CLINICAL TRIAL: NCT02300285
Title: Efficacy of Continuous Glucose Monitoring in Neonates With Hypoglycemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient eligible participants to meet recruitment goal
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Agus, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00014699
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hypoglycemia; Newborn Morbidity
MeSH Terms: conditions — Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGM Protocol (Experimental): Subjects will receive continuous glucose monitoring and caregivers will be able to view continuous glucose measurements.
  Interventions: Device: Continuous Glucose Monitoring
- Standard of Care (Placebo Comparator): Subjects will receive continuous glucose monitoring but caregivers will not be able to view continuous glucose measurements.
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Continuous glucose monitors (CGM) will be used to monitor blood sugar levels in enrolled subjects. CGMs measure blood sugar in the tissue just under the skin every few seconds and report average blood sugar every 5 minutes. In our study, the CGMs will function as monitoring systems. In the CGM protocol group the CGM will let the medical team know if there is a concerning blood sugar level, so that the medical team can then check a blood sugar level by the standard way (usually in a small drop of blood) and then decide if they need to give any medical treatment. In the Standard of Care group the CGM data will not be visible to the medical team but the medical team will be informed by the researchers if there are multiple unrecognized episodes of severe hypoglycemia.
  Other Names: Dexcom G4 Platinum

SUMMARY:
Our aim is to determine the feasibility of using continuous glucose monitors (CGMs) in infants with low blood glucose to improve how we care for these infants. To do this we plan on monitoring blood glucose levels with CGMs (instead of only with intermittent bloodsampling) in late-preterm and term infants admitted to the NICU who have had hypoglycemia. To see if using CGMs helps us prevent low blood glucose levels and allows us to find a diagnosis and treat sooner, we will randomize patients into one of two groups: a "CGM group" where the CGM information is made available to the NICU team and a "Standard of Care" group where the CGM information will only be available to the research team. However, if infants in the "Standard of Care" group are noted to have three unrecognized severe low blood glucose levels then the research team will inform the NICU team that this has occurred.

DETAILED DESCRIPTION:
We aim to evaluate the utility of continuous glucose monitors (CGMs) in improving the diagnosis and management of neonatal hypoglycemia in infants admitted to the neonatal intensive care unit (NICU). Specifically, we hope to assess whether the use of CGMs in this population reduces the number and severity of hypoglycemic events, reduces the time to diagnosis of the etiology of hypoglycemia and/or reduces the time taken to achieve stable euglycemia on a sustainable feeding regimen. We plan to perform a prospective pilot and feasibility study comparing the clinical course and outcomes of newborns with hypoglycemia admitted to the NICU who are actively monitored with CGMs versus those who receive routine care. Eligible infants will be late preterm and term infants admitted to the Boston Children's Hospital who have had two documented hypoglycemic episodes during their current admission. Families will be approached for consent shortly after diagnosis of recurrent hypoglycemia. As all of these infants will be undergoing periodic blood glucose monitoring as part of their routine care, enrollment in this study will involve minimal additional interventions, including CGM placement, which involves placement of a small subcutaneous needle sensor, and the possibility of drawing additional blood glucose samples if hypoglycemia is detected by CGM. All enrolled infants will be placed on a CGM monitor and then randomized to either the "CGM Protocol" or "Standard of Care" group. Those on the CGM Protocol will have a fully accessible CGM that will be analyzed for blood glucose trends and will alarm for any blood glucose level approaching hypoglycemic threshold (eg. BG <70 mg/dL). Those in the "Standard of Care" group will have a CGM in place, but values will not be available to the clinical team except if severe hypoglycemia is recorded (eg. BG <40 mg/dL). Whenever the CGM alarms or there is a concerning blood glucose trend as measured by the CGM, the nurse will be asked to check a blood glucose value. All clinical management decisions will be made by the clinical team based on confirmed blood glucose values. In the control group, the only change to current management is the potential performance of additional blood glucose checks that may be prompted by CGM alarms for severe hypoglycemia. The CGM will remain in place until the infant is no longer being monitored for glycemic stability or the infant is discharged. We will record all blood glucose levels, laboratory data related to investigation of the underlying cause of hypoglycemia, all intravenous and enteral sources of glucose, and uses of other therapeutic interventions such as diazoxide and carnitine replacement. We will also compare blood glucose data with information from the CGM monitors to assess accuracy. We will then compare severity and frequency of hypoglycemia, as well as times to diagnosis and euglycemia between the "CGM" and "Standard of Care" groups.

ELIGIBILITY:
Inclusion criteria:

* Age 0-60 days old
* Late-preterm and term infants (babies born more than 33 weeks and 6 days after the start of the pregnancy)
* History of low blood sugars (hypoglycemia): two episodes of hypoglycemia more than 1 hour apart (low blood sugar will be defined by age: for those less than 48 hours old a low blood sugar is considered less than 50mg/dL and for those older than 48 hours old less than 70mg/dL)

Exclusion Criteria:

* Infants with skin disease such that placement of a glucose sensor under the skin would be difficult to secure
* Infants expected to remain in NICU less than 24 hours
* Infants on a hypothermic protocol
* Infants enrolled in a competing clinical trial
* Family/team have decided to limit or redirect from aggressive NICU technological support
* infants who are wards of the state

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Steil GM, Langer M, Jaeger K, Alexander J, Gaies M, Agus MS. Value of continuous glucose monitoring for minimizing severe hypoglycemia during tight glycemic control. Pediatr Crit Care Med. 2011 Nov;12(6):643-8. doi: 10.1097/PCC.0b013e31821926a5. PMID 21499183
- [Background] Agus MS, Steil GM, Wypij D, Costello JM, Laussen PC, Langer M, Alexander JL, Scoppettuolo LA, Pigula FA, Charpie JR, Ohye RG, Gaies MG; SPECS Study Investigators. Tight glycemic control versus standard care after pediatric cardiac surgery. N Engl J Med. 2012 Sep 27;367(13):1208-19. doi: 10.1056/NEJMoa1206044. Epub 2012 Sep 7. PMID 22957521
- [Background] Agus MS, Asaro LA, Steil GM, Alexander JL, Silverman M, Wypij D, Gaies MG; SPECS Investigators. Tight glycemic control after pediatric cardiac surgery in high-risk patient populations: a secondary analysis of the safe pediatric euglycemia after cardiac surgery trial. Circulation. 2014 Jun 3;129(22):2297-304. doi: 10.1161/CIRCULATIONAHA.113.008124. Epub 2014 Mar 26. PMID 24671945

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Protocol: Subjects will receive continuous glucose monitoring and caregivers will be able to view continuous glucose measurements.
  Continuous Glucose Monitoring: Continuous glucose monitors (CGM) will be used to monitor blood sugar levels in enrolled subjects. CGMs measure blood sugar in the tissue just under the skin every few seconds and report average blood sugar every 5 minutes. In our study, the CGMs will function as monitoring systems. In the CGM protocol group the CGM will let the medical team know if there is a concerning blood sugar level, so that the medical team can then check a blood sugar level by the standard way (usually in a small drop of blood) and then decide if they need to give any medical treatment.
- Standard of Care: Subjects will receive continuous glucose monitoring but caregivers will not be able to view continuous glucose measurements.
  Continuous Glucose Monitoring: Continuous glucose monitors (CGM) will be used to monitor blood sugar levels in enrolled subjects. CGMs measure blood sugar in the tissue just under the skin every few seconds and report average blood sugar every 5 minutes. In our study, the CGMs will function as monitoring systems. In the Standard of Care group the CGM data will not be visible to the medical team but the medical team will be informed by the researchers if there are multiple unrecognized episodes of severe hypoglycemia.
Period: Overall Study
Arm/Group | CGM Protocol | Standard of Care
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Protocol | Standard of Care | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: Days] | 3.0 [2 to 5] | 3.33 [2 to 4] | 3.17 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hypoglycemic Events
Description: Hypoglycemia is defined by age group: for patients less than 48 hours of life, hypoglycemia is defined as glucose level < 50 mg/dL for patients greater than or equal to 48 hours of life it is defined as glucose level < 70 mg/dL.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | CGM Protocol | Standard of Care
Number analyzed (Participants) | 3 | 3
Events | 14 (2) | 19 (3)

2. Primary Outcome: Frequency of Severe Hypoglycemia Events
Description: Severe hypoglycemia is defined as glucose level < 40 mg/dL
Time Frame: Up to 28 days
Measure: Number; unit: Events
Arm/Group | CGM Protocol | Standard of Care
Number analyzed (Participants) | 3 | 3
Events | 1 | 4

3. Secondary Outcome: Number of Events Where Etiology of Hypoglycemia Was Established
Description: Diagnosis of the etiology of hypoglycemia, and the time to to do, will be evaluated in order to determine if the use of CGM will prompt earlier testing to evaluate the etiology of the hypoglycemia and therefore lead to earlier ascertainment of the underlying etiology. Diagnosis of etiology.
Time Frame: up tp 28 days
Population: Events of diagnosis of hyperinsulinemic hypoglycemia
Measure: Number; unit: Events
Arm/Group | CGM Protocol | Standard of Care
Number analyzed (Participants) | 3 | 3
Events | 2 | 1

4. Secondary Outcome: Time to Diagnosis of Etiology of Hypoglycemia
Description: Diagnosis of the etiology of hypoglycemia, and the time to to do, will be evaluated in order to determine if the use of CGM will prompt earlier testing to evaluate the etiology of the hypoglycemia and therefore lead to earlier ascertainment of the underlying etiology. Time to diagnosis of etiology.
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: Days
Arm/Group | CGM Protocol | Standard of Care
Number analyzed (Participants) | 3 | 3
Days | 1.5 [1 to 2] | 4 [4 to 4]

5. Secondary Outcome: Time to Stable Euglycemia
Time Frame: Up to 28 days
Population: Patients did not remain on protocol until euglycemia was reached, therefore no data was collected for this Outcome Measure.
Arm/Group | CGM Protocol | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days from enrollment and insertion of initial continuous glucose glucose monitor sensor.
Description: This is a Non-Significant-Risk (NSR) device study. If it is determined that an unanticipated adverse device effect presents an unreasonable risk to subjects, all investigations or parts of the investigations presenting that risk will be terminated as soon as possible and no later than 5 working days after the sponsor makes this determination. Because this is a small pilot study with minimal risk, no specific stopping rules will be developed and no interim analysis will be performed.
Arm/Group | CGM Protocol | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
The trial terminated due to lack of enrollment, thus limited data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02300285/Prot_SAP_000.pdf